CLINICAL TRIAL: NCT05160948
Title: Assessing Changes in Knowledge, Behavior, and Attitude Regarding Air Pollution After Receiving Personal Air Monitoring Results
Brief Title: Change in Knowledge After Receiving Personal Air Pollution Results
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2021-0707; 5R21ES030092-02 (NIH)
Record Dates: First submitted 2021-12-01; First posted 2021-12-16 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Environmental Exposure
Keywords: Ultrafine particle matter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Informational Report — All EcoMAPPE participants and their caregivers will be invited to complete a questionnaire to assess their understanding of air pollution and attitudes and beliefs about science and research before and after receiving their individual study air pollution monitoring results collected as part of their participation in EcoMAPPE.

SUMMARY:
Personal exposure to air pollution results from the interaction of individual time-activity patterns with levels of air pollution that vary over time and space. The increasing use of personal monitors capable of measuring geo-located and real-time air pollution in epidemiologic studies requires novel human subject considerations. Reporting individual exposure data back to participants is considered best practice in environmental health research using biomonitoring data and is beneficial to both study participants and researchers. The investigators believe that providing individual results of personal air monitoring may be more informative than biomonitoring data given the potential to increase participants' awareness of their exposure, identify specific locations and times of elevated exposures, and inform behavioral changes to decrease exposure and risk of adverse health outcomes.

DETAILED DESCRIPTION:
Personal exposure to air pollution results from the interaction of individual time-activity patterns with levels of air pollution that vary over time and space. Thus, personal monitors worn by study participants during daily living are considered the "gold-standard" to assess individual-level air pollution exposure. The increasing use of personal monitors capable of measuring geo-located and real-time air pollution in epidemiologic studies requires novel human subject considerations. In contrast with stationary air monitoring or models to estimate air pollution exposure, personal monitors provide a depth of insight and actionable information that is analogous to biological monitoring of chemical exposures. Reporting individual exposure data back to participants is considered best practice in environmental health research using biomonitoring data and is beneficial to both study participants and researchers. The investigators believe that providing individual results of personal air monitoring may be more informative than biomonitoring data given the potential to increase participants' awareness of their exposure, identify specific locations and times of elevated exposures, and inform behavioral changes to decrease exposure and risk of adverse health outcomes. Previously, the investigators enrolled adolescents in our Ecological Momentary Assessment and Personal Particle Exposure (EcoMAPPE) study (IRB #2017-1068) and measured personal exposure to ultrafine particles (UFPs; particulate matter <100 nm in diameter). Recently, the investigators conducted focus groups with a subset of EcoMAPPE participants (n = 16, IRB#: 2019-1003) with the purpose of co-designing information and report-back materials to provide study subjects' their individual results from personal sampling during their participation in the EcoMAPPE study. The overarching hypothesis of this current study is that providing EcoMAPPE participants and their caregivers with the results of their personal air pollution monitoring will increase their awareness and knowledge of their exposure to air pollution and strategies to reduce their exposure. The investigators propose one specific aim as part of this protocol: Aim 1: To increase study participants understanding of air pollution, associated health effects, and engagement with research. All EcoMAPPE participants and their caregivers will be invited to complete a questionnaire to assess their understanding of air pollution and attitudes and beliefs about science and research before and after receiving their individual study air pollution monitoring results collected as part of their participation in EcoMAPPE. All EcoMAPPE participants will be provided with their study results irrespective of their participation in this study.

The investigators will send an email invitation to caregivers of participants enrolled in the EcoMAPPE study. The investigators will also follow-up email invitations by phone call to provide additional information to EcoMAPPE participants and caregivers. Given that participants were ages 13-17 at enrollment, some EcoMAPPE participants are now adults (> 18 years of age) and the inestigators will also send an email invitation to participate to those participants. The email will contain information about the current study's objective and methods and a link to complete an electronic consent. The electronic consent will be completed by the participant (for those > 18) or their caregiver (for those < 18). The consent will specify that all EcoMAPPE participants and caregivers will receive their individual results irrespective of participating in this study. Following caregiver consent to participate in the study, participants will receive an invitation to participate and link to an electronic assent.

Following consent and assent, participants and their caregivers will each receive a "Report-Back Pre-Survey" via link to an electronic (Redcap) questionnaire. Participants and caregivers will complete the survey online via Redcap.

Following the completion of the "Report-Back Pre-Survey" caregivers and participants will receive an electronic (html) document containing the results of their EcoMAPPE participation. This report-back document contains information about the EcoMAPPE study, ultrafine particles, and the results of their individual personal sampling. The electronic (html) report-back document will be sent via Redcap.

After downloading and reviewing their personal report back document, participants and caregivers will receive a "Report-Back Post Survey" via link to an electronic REDCap questionnaire (attached). The "Report-Back Post Survey" will be similar to the "Report-Back Post Survey" and will ascertain changes in participants/caregivers attitudes and knowledge regarding air pollution and research.

If necessary (i.e. participant or parent does not have email), consenting and administration of study surveys will be done through an in person visit.

The investigators will compare changes in responses to questions on the Pre and Post Surveys using the paired t-test for questions answered on a 5-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have previously participated in the EcoMAPPE Study as a child or be a parent/legal guardian of a child that participated in EcoMAPPE

Exclusion Criteria:

- Not being a previous EcoMAPPE participant or parent of an EcoMAPPE participant

Ages: 15 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All EcoMAPPE participants and their caregivers will be invited to participate in this study. A total of 118 adolescents (age 13-17) were enrolled. Therefore, the sample size of this study is expected to be 236 (participant + caregiver). The sex and race of study participants is anticipated to reflect the enrollment in EcoMAPPE; 44% male, 74% White, 18% Black, and 8% other race.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Report-Back Pre/Post Survey | 12 months
  EcoMAPPE participants and their caregivers will be asked to complete a survey to assess their understanding of air pollution and beliefs about science and research before and after receiving their individual study monitoring results collected as part of their participation in EcoMAPPE. These questions will include Likert scale questions such as, 'On a scale from 1 to 5 (with 1 being 'very little' and 5 being 'a great deal), how much do you know about the health effects of air pollution?'). Other questions relate to how much participants know about the health effects of air pollution and air pollution sources. In addition to their personal monitoring data, the personalized reports will include basic information on particulate air pollution, sources, and reduction strategies.
  The investigators will compare their responses prior to reviewing their personalized report and their responses after reviewing their report to asses a shift in their awareness and knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ryan, PhD, Principal Investigator — CCHMC
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No